CLINICAL TRIAL: NCT06288308
Title: Fibrinogen to Albumin Ratio as a Predictive Biomarker for Lupus Nephritis (LN)
Brief Title: Fibrinogen to Albumin Ratio (FAR) as a Predictive Biomarker for Lupus Nephritis (LN)
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mamdouh Mohamed Fares, doctor, Assiut University
Other Study IDs: FAR in lupus nephritis (LN)
Record Dates: First submitted 2023-11-12; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fibronigin to albumin ratio — To investigate the association of fibrinogen to albumin ratio (FAR) with LN in different classes.
  b. Secondary (subsidiary):
  To prove the possible role of FAR as a novel diagnostic biomarker to predict LN progression

SUMMARY:
Fibrinogen to Albumin ratio as a predictive biomarker for lupus nephritis (LN)

DETAILED DESCRIPTION:
Systemic lupus erythematosus is a chronic autoimmune disease often coexists with other diseases and damages multiple organs such as kidney liver nervous system and so on.

Lupus nephritis is clinically evident in 50-60% of patients with systemic lupus erythematosus and it is histologically evident in most SLE patients even those without clinical manifestations of kidney disease .

The current standardized classification system for lupus nephritis is derived from the World Health Organization and the International Society of Nephrology/Renal Pathology Society's recommendations. The classification system is based on glomerular morphologic changes seen on microscopy immune deposits seen on immunofluorescence and also electronic microscopy.

Class 1 - Minimal Mesangial Lupus Nephritis. Class 2 - Mesangial Proliferative Lupus Nephritis. Class 3 - Focal Lupus Nephritis. Class 4 - Diffuse Lupus Nephritis. Class 5 - Membranous Lupus Nephritis. Class 6 - Advanced Sclerosis Lupus Nephritis. Fibrinogen (FIB) is an acute time response protein rises rapidly in inflammation infection myocardial infarction and tumor. The formation and deposition of immune complexes are important mechanism of lupus nephritis the infiltrate of inflammatory cells and the release of inflammatory factors cause renal injury resulting in the decreasing concentration of albumin. The fibrinogen-to-albumin ratio as a new inflammatory marker has been proved to have good predictive value in the diagnosis and prognosis of diabetic nephropathy acute renal injury SLE disease and so on.

ELIGIBILITY:
Inclusion Criteria:

1. 90 Pts with SLE that have LN in different classes.
2. Age between 18-60 yrs.

Exclusion Criteria:

1. Pts with ESRD, manifested cardiac valvular disease, acute infection, history of hepatitis, pts with DM and Cancer.
2. Age below 18 yrs& above 60 yrs
3. Pt who refused to contribute in this study

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Sample size was calculated using EPI info 2000 statistical package:- 60 patients diagnosed with LN depending on lab criteria and imaging are submitted for this study
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fibrinogen to Albumin ratio as a predictive biomarker for lupus nephritis (LN) | 1 year
  investigate the association of fibrinogen to albumin ratio (FAR) with LN and to prove its possible role as a novel biomarker to predict LN progression

REFERENCES:
- [Background] Parikh SV, Almaani S, Brodsky S, Rovin BH. Update on Lupus Nephritis: Core Curriculum 2020. Am J Kidney Dis. 2020 Aug;76(2):265-281. doi: 10.1053/j.ajkd.2019.10.017. Epub 2020 Mar 24. PMID 32220510
- [Background] Yap DYH, Chan TM. B Cell Abnormalities in Systemic Lupus Erythematosus and Lupus Nephritis-Role in Pathogenesis and Effect of Immunosuppressive Treatments. Int J Mol Sci. 2019 Dec 10;20(24):6231. doi: 10.3390/ijms20246231. PMID 31835612